CLINICAL TRIAL: NCT03991624
Title: Lack of Decision-making in Patients With Alzheimer's Disease : Functions Involved and the Daily Consequences
Acronym: MAPdP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 18CH237; 2019-A00174-53 (Other: ANSM)
Record Dates: First submitted 2019-02-25; First posted 2019-06-19 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Alzheimer Disease
Keywords: decision making; Iowa Gambling Task
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Alzheimer's patients (lack of executive functions) (Other)
  Interventions: Diagnostic Test: cognitive assessment; Other: Inhibition evaluation; Other: Assessment of mental flexibility; Other: Evaluation of the update
- control (lack of executive functions) (Other)
  Interventions: Diagnostic Test: cognitive assessment; Other: Inhibition evaluation; Other: Assessment of mental flexibility; Other: Evaluation of the update
- Alzheimer's patients (lack of working memory) (Other)
  Interventions: Diagnostic Test: cognitive assessment; Other: working memory
- control (lack of working memory) (Other)
  Interventions: Diagnostic Test: cognitive assessment; Other: working memory
- Alzheimer's patients (lack of episodic memory) (Other)
  Interventions: Diagnostic Test: cognitive assessment; Other: episodic memory
- control (lack of episodic memory) (Other)
  Interventions: Diagnostic Test: cognitive assessment; Other: episodic memory

INTERVENTIONS:
Diagnostic Test: cognitive assessment — * MMSE : Mini-Mental State Examination
  * 5 words of Dubois
  * Direct Assessment of Functional Status
  * Trail Making Test
  * BREF : Fast Front End Efficiency Battery
  * short battery of praxies
  * Quality of Life in Alzheimer's Disease
Other: Inhibition evaluation — * Stroop Victoria : This test consists of 3 sheets of 24 items, organized in 6 lines of 4 (points, neutral words or names of colours), from which the subject must identify the ink of the stimuli as quickly and precisely as possible.
  * Stop Signal task on the computer to give a response to the presentation of a target stimulus (Go signal) (e.g. pressing a button when a red circle appears on the screen, but doing nothing when a blue triangle appears), and prevent this response when the stimulus is followed or preceded by a beep (stop signal) (e.g. the appearance of a red circle is immediately preceded or followed by a beep, the subject should not press the button).
  Arms: Alzheimer's patients (lack of executive functions); control (lack of executive functions)
Other: Assessment of mental flexibility — * a letter-number pair task. The subject sees 4 blocks of 48 letter-number pairs appear successively on a screen. When the pair appears at the top, the subject must make a parity judgment but when the pair appears at the bottom, the subject must make a consonant / vowel judgment.
  * a category change task, which consists in classifying a word according to one category or another according to a visual clue that appears. The task consists of 4 blocks of 48 stimuli.
  Arms: Alzheimer's patients (lack of executive functions); control (lack of executive functions)
Other: Evaluation of the update — * an update span task for which letters appear on a screen sequentially, and subjects must memorize the last three, without knowing the length of the list. The task will consist of 3 tests of training and then 20 tests. After three errors consecutive, the task ends.
  * an n-back task that consists of a sequential presentation of letters, during which the subject must indicate when the stimulus. The task consists of 3 levels, with n = 1, n= 2 or n = 3. For level 1 (with n = 1), the subject must press a button when the same letter appears twice in a row on the screen. This task consists of 75 letters.
  Arms: Alzheimer's patients (lack of executive functions); control (lack of executive functions)
Other: working memory — * the empan baba task, which mainly involves maintaining information, and which consists in retaining a series of letters, appearing sequentially on a screen, and whose latency time between two word presentations is required for a secondary task: the repetition of baba syllables.
  * the task of reading operations which consists in recalling operations series of letters whose presentation is interspersed with the reading aloud of simple operations and of their results.
  * the ongoing operational task of recalling a list of letters, the presentation of which is interspersed with operations that are simple to read aloud and to to solve head-on.
  Arms: Alzheimer's patients (lack of working memory); control (lack of working memory)
Other: episodic memory — - A recognition task with a Remember/Know paradigm
  Arms: Alzheimer's patients (lack of episodic memory); control (lack of episodic memory)

SUMMARY:
Early in its development, Alzheimer's disease causes not only brain damage affecting different regions of the brain, such as the entorhinal cortex, the anterior cingulate cortex, and the prefrontal lobe, but also a cognitive deficit affecting several functions, such as episodic memory, executive functions, or working memory. Although these different areas and functions are involved in the decision-making process, few studies have focused their research on this subject in the context of Alzheimer's disease. However, a 2008 study showed an early decline in decision-making skills in the disease, but did not link this deficit to cognitive impairment. In addition, decision-making is generally assessed using a test called the Iowa Gambling Task (IGT), which, despite its many advantages, does not have established ecological validity.

In the context of pathology, however, it seems essential to evaluate decision-making in relation to daily life, especially since a deficit in this process would have considerable repercussions on quality of life.

In this study, the investigators seek to better define the disorder by decision-making in early Alzheimer's disease, to understand the links between them with the deficit of other cognitive functions, and to highlight the the consequences that this decline has on patients' daily lives.

ELIGIBILITY:
Inclusion Criteria for patients with Alzheimer's disease :

* Mini-Mental State Examination > 23
* stable treatment for at least two months
* mother tongue : French

Inclusion Criteria for control :

* general cognitive level in the standard on the following tests : Mini-Mental State Examination and Fast Front End Efficiency Battery
* mother tongue : French

Exclusion Criteria for patients with Alzheimer's disease :

* game addiction
* uncorrected visual and hearing disorders
* other neurological or psychiatric history
* inability to communicate
* delusional or psychotic state

Exclusion Criteria for control :

* game addiction
* psychiatric or neurological disorders
* anxiety and depression symptomatology

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2019-09-27 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Score obtained (the number of correct answers) by participants in tasks evaluating decision-making | day 14
  measured with two decision-making tasks : Iowa Gambling Task and one experimental task

SECONDARY OUTCOMES:
Score obtained in task evaluating executive functions | day 14
  measured with Stroop Victoria
Score obtained in task evaluating executive functions | day 14
  measured with Stop Signal on computer
Score obtained in task evaluating executive functions | day 14
  measured with a letter-number pair task
Score obtained in task evaluating executive functions | day 14
  measured with a category change task.
Score obtained in task evaluating executive functions | day 14
  measured with an update span task and a n-back task.
Score obtained in task evaluating working memory | day 14
  measured with the task of empan baba.
Score obtained in task evaluating working memory | day 14
  measured with the task of reading operations.
Score obtained in task evaluating working memory | day 14
  measured with the continuous operation task.
Scores obtained in tasks evaluating episodic memory | day 14
  measured with a recognition task with a Remember/Know paradigm
Scores obtained from the quality of life questionnaire. | day 14
  measured with Quality of Life in Alzheimer's Disease : it is composed of 13 items (ex: physical health, memory, relationship with friends...). the patient must rate according to 4 possibilities: bad, fairly good, good or excellent. There is one copy to be completed by the patient and another by the caregiver.
Scores obtained from autonomy questionnaire. | day 14
  measured with Direct Assessment of Functional Status : assessment of several areas of daily life (spatial and temporal orientation, communication skills, driving, financial management, shopping ability, behaviour food and hygiene). It consists of 7 subscales, allowing each competency to be assessed independently.

CONTACTS AND LOCATIONS:
Overall Officials: Céline BORG, Principal Investigator — CHU de Saint Etienne
Locations (4):
- France (4):
  - Laboratoire d'Etude des Mécanismes Cognitifs, Bron
  - Hôpital Lariboisière- Fernand Widal, Paris
  - CHU de Saint Etienne, Saint-Etienne
  - CMRR - Hôpital Charpennes, Villeurbanne

IPD SHARING:
Plan to Share IPD: No